CLINICAL TRIAL: NCT00987350
Title: A Clinical Study to Assess the Safety, Tolerability, and Immunogenicity of Licensed Seasonal Trivalent Influenza Vaccine Administered by Needle-free Jet Injection in One Intramuscular Dose to Healthy Young Adults
Brief Title: Safety Study of Seasonal Influenza Vaccine by Jet Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: D'Antonio Consultants International, Inc. (Other)
Responsible Party: Principal Investigator, Karen Kotloff, Division Head, Ped-Infectious Diseases and Tropical Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: HP-00042669; LectraJet-TIV CVD 1000
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy Adults
Keywords: Jet Injector; Vaccine; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trivalent influenza vaccine by needle and syringe (Active Comparator): Thirty volunteers will receive 1 intramuscular (IM) dose of licensed trivalent inactivated 2009-10 seasonal influenza vaccine by the standard needle and syringe method
  Interventions: Device: TIV by jet injection; Biological: Seasonal Trivalent Influenza Vaccine
- Trivalent influenza vaccine by jet injection (Experimental): Thirty volunteers will receive 1 intramuscular (IM) dose of licensed trivalent inactivated 2009-10 seasonal influenza vaccine by the experimental method of jet injection
  Interventions: Device: LectraJet; Biological: Seasonal Trivalent Influenza Vaccine

INTERVENTIONS:
Device: LectraJet — LectraJet is a new jet injector studied for the first time in humans. It is in the category known as disposable-syringe jet injectors that have the advantage of eliminating the risk of disease transmission between subjects. A new syringe and nozzle is used for each patient so that no splash back of blood can occur onto the jet apparatus itself.
  Arms: Trivalent influenza vaccine by jet injection
Device: TIV by jet injection — Administration of seasonal trivalent influenza vaccine (TIV) by jet injection
  Arms: Trivalent influenza vaccine by needle and syringe
Biological: Seasonal Trivalent Influenza Vaccine — Licensed trivalent influenza vaccine provided by either jet injection or traditional needle and syringe.

SUMMARY:
This research study involves testing of a device that can give injections (shots) without the use of a needle.

DETAILED DESCRIPTION:
The device is called LectraJet M3 and has recently been approved by the Food and Drug Administration (or FDA), the government agency that oversees the approval of new medical devices. The approval is called a 510(k) and allows for the marketing and use of the device in the United States (US). Devices under a 510(k) do not need to have clinical trials performed. The researchers are performing this study in order to collect clinical data in a controlled environment. Non significant risk (NSR) devices such as the LectraJet may be studied in clinical trials with or without a 510(k). Currently there are several other disposable-syringe jet injectors that are also FDA approved for sale and use in the United States, including: 1) Biojector® 2000 , 2) Medi-Jector Vision, and 3) Injex™. These devices have been used to deliver millions of injections in a variety of healthcare settings. The LectraJet® is jet injector that is most suited for mass immunization campaigns due to the ability to power the device with a foot pedal as well as electricity and the speed with which immunizations can be delivered. It is designed so that vaccine delivery characteristics are the same as that of the licensed disposable-syringe jet injectors.

Giving vaccines without needles (needle-free vaccine delivery) may be better than giving them using a needle for many reasons. One method for giving shots without needles is a technique called jet injection. This is what the researchers are testing in this study. A jet injector pushes the vaccine fluid out of a small hole at a high enough speed to allow the vaccine to go under the subject's skin without needing a needle. Years ago, people got shots using jet injectors, but these older devices reused the same "nozzle" or hole through which the fluid was forced. Newer jet injectors, including the one the researchers are testing in this study, use disposable cartridges to hold the vaccine. So, the only thing that touches the subject's skin is their own cartridge, which gets thrown away after injection.

In this study, the volunteers are getting the licensed seasonal flu vaccine to see if the jet injector works as well as giving the vaccine by needle and syringe. The seasonal flu vaccine that the researchers are using is called trivalent influenza vaccine (TIV). It is licensed in the US to protect people 6 months of age and older against influenza. Influenza is a virus that is also commonly known as the "flu". The flu is a serious illness that kills over 35,000 people per year in the US alone. The flu virus constantly changes and that is why people who are at risk for developing complications from the flu, such as children, the elderly, and people with underlying health conditions need to be vaccinated every year. Volunteers will receive the 2009-2010 annual seasonal flu vaccine called TIV either by needle and syringe or by jet injection. The researchers will compare the side effects and see how well the vaccine generates an immune response when given by the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and 49 years, inclusive
* In good health as evidenced by screening evaluation within the 30 days prior to immunization.
* Expressed interest and availability to fulfill the study requirements.
* Signed, informed consent.
* For women of child-bearing potential, agreement to avoid pregnancy for the 90 days following vaccination by use of effective birth control methods.
* Agreement to refrain from taking any experimental drug or vaccine from Day minus 30 to Day 90 (from screening until the volunteer completes the study).

Exclusion Criteria:

* A known allergy to a component of the vaccine, including egg, egg products, chicken proteins, formaldehyde, gentamicin sulfate, or sodium deoxycholate.
* A positive urine pregnancy test in the 24 hours prior to vaccination. (A negative urine pregnancy test is required within the 24 before vaccination for all women who have not had a hysterectomy or are not at least 1 year post-menopausal)
* A woman who is breastfeeding.
* Any current medical illness that might jeopardize the volunteer's safety or interfere with the interpretation of the study results. These include, but are not limited to the following: cancer; immunodeficiency; bleeding disorder.
* Any underlying medical condition for which influenza vaccination is recommended: chronic heart or lung conditions, including asthma; metabolic diseases; kidney disease; blood disorder (such as sickle cell anemia); weakened immune systems, including HIV/AIDS.
* Resident of nursing homes and long term care facility.
* Health care worker involved in direct patient care.
* Any current illness requiring daily medication, except for vitamins, contraceptives, topical medications, antihistamines, antacids and other reflux medications, smoking cessation medications, headache medications that do not have antipyretic activity, nasal allergy medications, ophthalmologic and otic medications, psychiatric medications for well-controlled conditions such as depression or anxiety, and thyroxine for stable, inactive hypothyroidism. Volunteers may not take daily oral, nasal, inhaled, or parenteral steroids or non-steroidal anti-inflammatory medications. Medications other than those mentioned above will require approval from the PI, the sponsor, and the medical monitor.
* Any use of antibiotics in the 7 days before enrollment.
* Vital signs that are abnormal and thought by the investigator to increase the risk to the volunteer. Mild elevations or depressions of blood pressure or heart rate may be allowed.
* Current alcohol or illicit drug dependence.
* History of receipt of an influenza vaccine in the 2008-2009 and/or 2009-2010 season
* History of Guillain-Barré Syndrome
* Failure to pass the written exam; a passing score is 70% or greater.
* Receipt of an experimental agent (e.g., a vaccine or medication) within the 30 days prior to enrollment or the expectation of receipt of an experimental agent while participating in this study.
* Receipt of a live, attenuated vaccine within the 30 days prior to enrollment.
* Receipt of a subunit or killed vaccine within the 14 days prior to enrollment.
* Receipt of a blood product, including immunoglobulin, in the 90 days prior to enrollment.
* Oral temperature > 37.7 degrees C or other acute illness occurring prior to inoculation on the day of vaccination. (This will lead to postponement of enrollment, not exclusion from the trial. Mild resolving illnesses may be allowed at the discretion of the investigator)
* Anything that, in the opinion of the investigator, will compromise the participation of the volunteer with respect to his/her rights or risks.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) and serious adverse event (SAE) information (solicited in the clinic and via memory aids, concomitant medications, and periodic targeted physical assessment) | 90 Days

SECONDARY OUTCOMES:
Proportion of volunteers in each administration group achieving a greater than four-fold rise in hemagglutination inhibition (HI) titer from pre-vaccination to 28 days post-vaccination against each of the vaccine-associated strains | Day 28
Proportion of volunteers in each administration group achieving a HI titer >40 on day 28 post-vaccination against each of the vaccine-associated strains | Day 28
Geometric mean titer (GMT) of HI titers against each of the vaccine-associated strains in each group 28 days after receipt of the vaccine | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jakub K Simon, MD, MS, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland College Park Health Center, College Park, Maryland, United States

REFERENCES:
- [Background] Parent du Chatelet I, Lang J, Schlumberger M, Vidor E, Soula G, Genet A, Standaert SM, Saliou P. Clinical immunogenicity and tolerance studies of liquid vaccines delivered by jet-injector and a new single-use cartridge (Imule): comparison with standard syringe injection. Imule Investigators Group. Vaccine. 1997 Mar;15(4):449-58. doi: 10.1016/s0264-410x(96)00173-9. PMID 9141217
- [Background] Fisch A, Cadilhac P, Vidor E, Prazuck T, Dublanchet A, Lafaix C. Immunogenicity and safety of a new inactivated hepatitis A vaccine: a clinical trial with comparison of administration route. Vaccine. 1996 Aug;14(12):1132-6. doi: 10.1016/0264-410x(96)00044-8. PMID 8911009
- [Background] Williams J, Fox-Leyva L, Christensen C, Fisher D, Schlicting E, Snowball M, Negus S, Mayers J, Koller R, Stout R. Hepatitis A vaccine administration: comparison between jet-injector and needle injection. Vaccine. 2000 Mar 17;18(18):1939-43. doi: 10.1016/s0264-410x(99)00446-6. PMID 10699344